CLINICAL TRIAL: NCT05185869
Title: A Phase II Study of SHR6390 Plus Nab-paclitaxel and Gemcitabine in Unresectable Advanced/Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: SHR6390 Plus Nab-paclitaxel and Gemcitabine in Advanced/Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC-1st-IIT-SHR6390-AG
Record Dates: First submitted 2021-12-19; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AG+SHR6390 (Experimental): Subjects will receive SHR6390 plus nab-paclitaxel and gemcitabine
  Interventions: Drug: SHR6390; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: SHR6390 — SHR6390, Oral Administration
Drug: Nab-paclitaxel — Paclitaxel-albumin, Intravenous Injection
Drug: Gemcitabine — Gemcitabine, Intravenous Injection

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of SHR6390 in combination with nab-paclitaxel and gemcitabine in first-line treatment of subjects with advanced/metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is an open-label, prospective, single-center, single-arm, Simon's two-stage design phase II study for unresectable advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) subjects treated with SHR6390 plus nab-paclitaxel and gemcitabine.

In this research study, the main objectives include:

1. Evaluate objective response rate in patients with pancreatic cancer receiving SHR6390 plus nab-paclitaxel and gemcitabine.
2. Assess adverse side effects associated with the combination of SHR6390 with nab-paclitaxel and gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of 18 to 75 years old;
2. Subjects are diagnosed with histologically confirmed unresectable advanced or metastatic pancreatic ductal adenocarcinoma with at least one measurable lesion according to the RECIST 1.1 standard (the CT scan length of the tumor lesion > 10 mm);
3. Subjects are naïve to systemic treatment;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
5. Life expectancy ≥12 weeks;
6. Adequate organ performance based on laboratory blood tests;
7. The toxicity of the previous treatment has been restored to ≤1 level (if there is surgery, the wound has completely healed);
8. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation;
9. Normal swallowing function;
10. Willing to consent and signed the informed consent, and able comply with the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

1. Had other active malignant tumors within 5 years before entering the study;
2. Confirmed or suspicious new metastatic lesion in brain;
3. Subjects are allergy to experimental drugs or any excipients;
4. Coagulation disorders (INR>1.5, APTT>ULN);
5. Severe pleural effusion or ascites;
6. Severe and uncontrolled medical diseases, acute infections; recent history of major surgery for myocardial infarction (within 3 months);
7. Subjects combined with other anti-tumor drugs;
8. Chronic diarrhea or intestinal obstruction;
9. Pregnant or lactating women; Fertile subjects who are unwilling or unable to take effective contraceptive measures;
10. Subjects in any trial drug treatment;
11. Severe mental disorder;
12. Other situations that investigators considered should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years.
  ORR is defined as the proportion of patients with best objective response of confirmed complete response (CR) or partial response (PR) according to RECIST1.1.
Adverse Events (AEs) | From the first drugs administration to within 30 days for the last treatment.
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 2 years.
  OS is defined as the time from the first drugs administration to the date of death due to any cause or the last follow ship.
Progression Free Survival (PFS) | Up to 2 years.
  PFS is defined as the time from the first drugs administration to the date of disease progression or the last follow ship.
Disease Control Rate (DCR) | Up to 2 years.
  DCR is defined as the rate of participants who have achieved complete response, partial response and stable disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No